CLINICAL TRIAL: NCT03198507
Title: A Randomized Double Blind Active Comparator Controlled Phase III Study to Assess the Safety and Efficacy of RHB-105 in the Treatment of Confirmed Helicobacter Pylori (H. Pylori) Infection
Brief Title: ERADICATE Hp2 - Treating Helicobacter Pylori With RHB-105 Compared to Active Comparator
Acronym: ERADICATE Hp2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RedHill Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RHB-105-02
Record Dates: First submitted 2017-06-07; First posted 2017-06-26 (Actual); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2018-08

CONDITIONS: Helicobacter Pylori Infection; Dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — Amoxicillin; Omeprazole; Rifabutin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RHB-105 (Experimental): RHB-105 is an 'all-in-one' combination oral capsule consisting of combination therapy of Amoxicillin, Omeprazole and Rifabutin; as well as separate Riboflavin
  Interventions: Drug: RHB-105
- Active Comparator (Active Comparator): Active comparator is an 'all-in-one' combination oral capsule consisting of combination therapy of Amoxicillin and Omeprazole; as well as separate Riboflavin
  Interventions: Drug: Active Comparator

INTERVENTIONS:
Drug: RHB-105 — The intended dose of RHB-105 (12.5 mg rifabutin, 250 mg amoxicillin, and 10 mg omeprazole capsules) 4 capsules every eight hours, is equivalent to a total daily dose of:
  * Rifabutin 150 mg
  * Amoxicillin 3000 mg
  * Omeprazole 120 mg
  One 50mg Riboflavin tablet to be taken once daily to maintain the blind.
  Other Names: Amoxicillin, Omeprazole and Rifabutin
  Arms: RHB-105
Drug: Active Comparator — The intended dose of the Active Comparator (250 mg amoxicillin, and 10 mg omeprazole capsules) 4 capsules every eight hours, equivalent to a total daily dose of:
  * Amoxicillin 3000 mg
  * Omeprazole 120 mg
  One 50mg Riboflavin tablet to be taken once daily to maintain the blind.
  Other Names: Amoxicillin and Omeprazole
  Arms: Active Comparator

SUMMARY:
The "test and treat" strategy for treating dyspeptic patients who are H. pylori positive is rapidly becoming the standard of care. This study will test the effectiveness of RHB-105, a new triple therapy to treat H. pylori infection in dyspeptic patients against an active comparator.

DETAILED DESCRIPTION:
This is a, randomized, double blind, active comparator-controlled study of RHB-105 in adult subjects complaining of epigastric discomfort that have been screened and found to be positive for H. pylori infection via 13C UBT and gastric biopsy.

The biopsy samples will also be used to conduct H. pylori antibiotic susceptibility/resistance assessment.

The study will be conducted at up to 65 sites in the USA. Eligible subjects will be randomized in a ratio of 1:1 between the RHB-105 arm (n=222) and the active comparator arm (n=222). Subjects will receive RHB-105 or active comparator for 14 consecutive days. Eradication of H. pylori infection will be determined at Visit 5 based on 13C UBT testing conducted between 43 and 71 days after initiation of study drug therapy.

All subjects who meet inclusion and exclusion criteria and have positive13C UBT will undergo upper endoscopy with sampling for culture and sensitivity testing (to rifabutin, amoxicillin, clarithromycin, and metronidazole) prior to randomization. After test of cure at Visit 5, all H. pylori eradication failures will receive susceptibility directed Standard of Care therapy based on initial culture results for subjects, and undergo repeat upper endoscopy for post treatment antibiotic susceptibility/resistance assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Be ages 18 - 70, inclusive; non-Asian males and females (This population has been demonstrated to have significantly elevated omeprazole levels as per the prescriber information for other omeprazole products). A person having origins in any of the original peoples of the Far East, Southeast Asia, or the Indian subcontinent, including, for example, Cambodia, China, India, Japan, Korea, Malaysia, Pakistan, the Philippine Islands, Thailand, and Vietnam should be considered Asian, and forr this study Asian is defined as having at least one Asian grandparent (Shektar et al, 2014, FDA Guidance for Industry 2016);
2. Positive for H. pylori by 13C Urea Breath Test (UBT) and confirmed positive via gastric biopsy for campylobacter-like organism (CLO) Rapid Urease Test, or H. pylori culture or histology;
3. Symptoms consistent with dyspepsia of at least two weeks duration (defined as recurrent pain or discomfort centered in the upper abdomen, often with a relation to meals);
4. Females must not be pregnant or lactating and:

   1. at no risk of pregnancy for one of the following reasons: postmenopausal for at least one year from the date of informed consent, status post hysterectomy or tubal ligation, OR
   2. are prepared to and agree to use of an intrauterine device (IUD) or practice double method birth control (barrier plus spermicide) from screening through to 30 days post-end of-treatment (EOT); Acceptable double contraceptive methods include barrier (condoms or diaphragms) plus spermicide
   3. Hormonal contraceptives (birth control pills and hormone implants) are not acceptable contraception methods under this protocol;
5. Males must be surgically sterilized or are prepared to and agree to practice double method (barrier plus spermicide) birth control from screening through to 30 days post-EOT;
6. Agree to refrain from consuming alcohol from 1 week prior to screening to Test of Cure/Visit 5;
7. Agree to refrain from taking antacids from screening through day 15 and for at least 24 hours prior to Test of Cure/Visit 5 and if applicable at least 24 hours prior to Visit 8/Test of Cure;
8. Agree to refrain from taking H2 blockers at least 24 hours prior to screening 13C UBT and at least 24 hours prior to Test of Cure/Visit 5 and if applicable at least 24 hours prior to Visit 8/Test of Cure;
9. Agree to refrain from taking sucralfate from one week prior to screening through Test of Cure/Visit5;
10. Agree to refrain from taking bismuth containing medications such as Pepto-BismolTM or other proton pump inhibitors (PPIs) from two weeks prior to screening through Test of Cure/Visit 5;
11. Agrees to refrain from consuming grapefruit, or any other food or supplement known to significantly affect CYP3A4 or CYP2C19 activity from screening to day 15;
12. Provide written informed consent to participate as shown by a signature of subject on the consent form.

Exclusion Criteria:

1. Have alarm symptoms/signs (including unexplained anemia [iron deficiency], melena / hematemesis, anorexia, dysphagia, jaundice, weight loss);
2. Have received prior H. pylori eradication therapy;
3. Use of antibiotics in the 4 weeks immediately prior to screening 13C UBT;
4. Use of any proton pump inhibitors (PPIs) or bismuth-containing medications (such as Pepto-BismolTM) within the 2 weeks immediately prior to screening 13C UBT;
5. Use of any of the following medications within seven days prior screening: alfentanil, allopurinol, amlodipine, anti-herpes agents, anti-retroviral agents, apixaban, aprepitant, aripiprazole, astemizole, atorvastatin, boceprevir, buspirone, carbamazepine, cisapride, citalopram dosed greater than 20 mg /d, clomipramine, clopidogrel and other oral anticoagulants, colchicine, dapsone, dihydroergotamine, digoxin, diltiazem, ergotamine, felodipine, fluconazole, gleevec, hormonal contraceptives that are not exclusively norethindrone or norgestrel, imipramine, itraconazole, ketoconazole, latuda, lovastatin, mycophenolate mofetil, nifedipine, nisoldipine, nitrendipine, phenytoin, pimozide, probenecid, proguanil, quinine, roflumilast, terfenadine and voriconazole;
6. Use of amiodarone;
7. Presence of more than two active gastric and/or duodenal ulcers;
8. History of gastric outlet obstruction; or hypersecretory state (e.g., Zollinger Ellison Syndrome);
9. History of esophageal or gastric surgery, except for simple closure of perforated ulcer;
10. History of gastric cancer;
11. History of malignancy within the past five years except for basal cell carcinoma of the skin or carcinoma in situ of the cervix that has been treated with no evidence of recurrence;
12. Positive screening laboratory results for human immunodeficiency virus (HIV) antibody (HIV1 or HIV2), or hepatitis B surface antigen (HBs Ag), or hepatitis C antibody (HCV Ab), unless patient has documented sustained viral response evidenced by prior and/or current absence of viral RNA at least 24 weeks after completing antiviral therapy;
13. Current drug or alcohol abuse or history of drug or alcohol abuse in the past 5 years from screening;
14. Known hypersensitivity or suspected history of hypersensitivity reactions to any of the study drugs or related drugs, including cephalosporins and penicillin;
15. Clinical evidence of any disease that in the opinion of the investigator might interfere with the subject's ability to participate in the trial;
16. History of QT prolongation (QTc greater than 450ms in males and 460ms in females), or ventricular arrhythmia, including torsades de pointes;
17. Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) >3x Upper Limit of Normal (ULN), or Alkaline Phosphatase (APO4) >2x ULN, or Total Bilirubin >2x ULN. Subjects with confirmed diagnosis of Gilbert's Syndrome are excluded if Total Bilirubin > 2.5x ULN;
18. Unable to communicate well with the Investigators and to comply with the study requirements;
19. Involved in any other experimental drug or device protocol (outside of this RHB-105-02 study) within the 4 weeks immediately prior to screening visit through end of study;
20. Subjects with creatinine clearance less than 30 ml/min at screening via estimated Cockcroft-Gault (eCGF) formula: eCGF or estimated creatinine clearance = [140 - age in years] * weight (kg) / 72 * Serum Creatinine (mg/dl) [multiply estimated rate by 0.85 for women], using actual body weight at screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2017-06-18 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Graham, MD, Principal Investigator — Baylor College of Medicine
Locations (51):
- United States (51):
  - Research Site, Dothan, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, North Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Chula Vista, California
  - Research Site, Lomita, California
  - Research site, San Carlos, California
  - Research Site, Bristol, Connecticut
  - Research Site, Aventura, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Homestead, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Miami, Florida
  - Research Site, Orange City, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Athens, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Elwood, Indiana
  - Research Site, Metairie, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Chevy Chase, Maryland
  - Research Site, Brockton, Massachusetts
  - Research Site, Chesterfield, Missouri
  - Research Site, Wyoming, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Great Neck, New York
  - Research Site, Concord, North Carolina
  - Research Site, Davidson, North Carolina
  - Research Site, Fayetteville, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Tulsa, Oklahoma
  - Research Site, Greenville, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research site, Hermitage, Tennessee
  - Research Site, Nashville, Tennessee
  - Research site, Houston, Texas
  - Research Site, Houston, Texas
  - Research Center, Houston, Texas
  - Research Site, Longview, Texas
  - Research Site, Richardson, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Ogden, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Christiansburg, Virginia
  - Research Site, Lynchburg, Virginia
  - Research site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Howden CW, Sheldon KL, Almenoff JS, Chey WD. Pitfalls of Physician-Directed Treatment of Helicobacter pylori: Results from Two Phase 3 Clinical Trials and Real-World Prescribing Data. Dig Dis Sci. 2022 Sep;67(9):4382-4386. doi: 10.1007/s10620-021-07323-5. Epub 2021 Dec 4. PMID 34862940
- [Derived] Graham DY, Canaan Y, Maher J, Wiener G, Hulten KG, Kalfus IN. Rifabutin-Based Triple Therapy (RHB-105) for Helicobacter pylori Eradication: A Double-Blind, Randomized, Controlled Trial. Ann Intern Med. 2020 Jun 16;172(12):795-802. doi: 10.7326/M19-3734. Epub 2020 May 5. PMID 32365359

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between July 2017 and December 2018. A total of 62 centers in the US screened potential subjects and 55 centers randomized subjects into the study.
Groups:
- RHB-105: RHB-105 (Rifabutin 150 mg, Amoxicillin 3000 mg, Omeprazole 120 mg)
- Active Comparator: Active comparator (Amoxicillin 3000 mg, Omeprazole 120 mg)
Period: Overall Study
Arm/Group | RHB-105 | Active Comparator
Started | 228 | 227
Completed | 227 | 227
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treatment naïve adult subjects aged 18 to 70 years, complaining of epigastric discomfort that had been screened and found to be positive for H. pylori infection via 13C UBT and follow up upper endoscopy (culture, histology, or CLO test).
Groups:
- Total: Total of all reporting groups
Arm/Group | RHB-105 | Active Comparator | Total
Number analyzed (Participants) | 228 | 227 | 455
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 214 | 207 | 421
  >=65 years | 14 | 20 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (12.77) | 47.2 (13.13) | 46.5 (12.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 151 | 283
  Male | 96 | 76 | 172
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 149 | 124 | 273
  Not Hispanic or Latino | 79 | 103 | 182
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 3 | 3
  Race: Asian | 0 | 0 | 0
  Race: Black or African American | 35 | 53 | 88
  Race: Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Race: White | 184 | 167 | 351
  Race: Other | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 228 | 227 | 455
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 30.32 (6.027) | 30.95 (6.886) | 30.63 (6.470)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Eradication of H. Pylori
Description: Eradication of H. pylori confirmed via 13C Urea Breath Test (UBT) testing. Subjects with negative test results (eradication of H. pylori) were considered treatment successes. Subjects who tested positive for H. pylori infection (no eradication) were considered treatment failures.
Time Frame: 43-71 days after initiation of treatment
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-105 | Active Comparator
Number analyzed (Participants) | 228 | 227
Participants | 191 | 131
Statistical Analysis 1: Comparison: RHB-105 vs Active Comparator; Test type: Superiority; p = 0.0001, t-test, 2 sided — Statistical testing was 2 sided and performed using a significance (alpha) level of 0.05

2. Secondary Outcome: Number of Participants With H. Pylori Cultures That Presented Antibiotic Resistance and Susceptibility
Description: The primary endpoint was summarized within subgroups formed by the presence of H. pylori susceptibility and resistance to amoxicillin, clarithromycin, metronidazole, and rifabutin from H. pylori cultures from samples obtained prior to initiating study treatment (i.e. baseline).
  A participant is considered a responder when H. pylori is eradicated after treatment as confirmed via 13C Urea Breath Test (UBT). A participant is considered a non-responder when H. pylori is not eradicated after treatment.
Time Frame: 43-71 days after initiation of treatment
Population: n is the number of cultures obtained from the in the FAS population in each treatment group with H. pylori resistant/susceptible to Rifabutin, Amoxicillin, Clarithromycin or Metronidazole at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-105 | Active Comparator
Number analyzed (Participants) | 174 | 171
Participants
  Rifabutin resistant: number analyzed (Participants) | 0 | 0
  Rifabutin resistant: Responder | 0 | 0
  Rifabutin resistant: Non-responder | 0 | 0
  Rifabutin Susceptible: Responder | 147 | 99
  Rifabutin Susceptible: Non-responder | 27 | 72
  Amoxicillin Resistant: number analyzed (Participants) | 13 | 9
  Amoxicillin Resistant: Responder | 9 | 4
  Amoxicillin Resistant: Non-responder | 4 | 5
  Amoxicillin Susceptible: number analyzed (Participants) | 161 | 162
  Amoxicillin Susceptible: Responder | 138 | 95
  Amoxicillin Susceptible: Non-responder | 23 | 67
  Clarithromycin Resistant: number analyzed (Participants) | 25 | 35
  Clarithromycin Resistant: Responder | 21 | 22
  Clarithromycin Resistant: Non-responder | 4 | 13
  Clarithromycin Susceptible: number analyzed (Participants) | 149 | 136
  Clarithromycin Susceptible: Responder | 126 | 77
  Clarithromycin Susceptible: Non-responder | 23 | 59
  Metronidazole Resistant: number analyzed (Participants) | 71 | 79
  Metronidazole Resistant: Responder | 57 | 45
  Metronidazole Resistant: Non-responder | 14 | 34
  Metronidazole Susceptible: number analyzed (Participants) | 103 | 91
  Metronidazole Susceptible: Responder | 90 | 53
  Metronidazole Susceptible: Non-responder | 13 | 38

3. Secondary Outcome: Number of Participants With Adverse Events That Are Related to Treatment
Description: The number of participants that presented treatment emergent adverse events (TEAE) during the study overall, TEAEs related to study drug and severe TEAEs.
Time Frame: After first dose of study drug until 28 days following last dose.
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-105 | Active Comparator
Number analyzed (Participants) | 228 | 227
Participants
  No. of subjects with any TEAE | 83 | 72
  No. of subjects with any study drug related TEAE | 47 | 44
  No. of subjects with any severe TEAE | 4 | 4

4. Other Pre Specified Outcome: Number of Participants With Eradication of H. Pylori in the Pharmacokinetic Population (PKP)
Description: A pre-specified responder analysis of eradication of H. pylori confirmed via 13C Urea Breath Test (UBT) was performed in the PK population.
  The PK population was generated based on the measurement of plasma concentrations of amoxicillin, omeprazole, rifabutin, and the rifabutin metabolite 25-O-desacetyl-rifabutin (on Day 13). It included those subjects in the FAS who had demonstrable presence of any component of investigational drug at Visit 3 or had no levels detected >250 hours after the last dose. For all subjects, the reason for exclusion from the PKP was the absence of any pharmacokinetic component of study drug at Visit 3 within 250 hours of the last reported dose. Two hundred fifty hours was selected to account for approximately 10 times the terminal half-life of rifabutin.
Time Frame: 43-71 days after initiation of treatment
Population: Pharmacokinetic Population (PKP)
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-105 | Active Comparator
Number analyzed (Participants) | 207 | 184
Participants | 187 | 119
Statistical Analysis 1: Comparison: RHB-105 vs Active Comparator; Test type: Superiority; p = 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events reported from first study drug administration and until 28 days following the last dose of blinded study drug.
Arm/Group | RHB-105 | Active Comparator
All-Cause Mortality (participants affected / at risk) | 0/228 | 0/227
Serious Adverse Events (participants affected / at risk) | 1/228 | 1/227
Other Adverse Events (participants affected / at risk) | 51/228 | 46/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RHB-105 (N=228) | Active Comparator (N=227)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RHB-105 (N=228) | Active Comparator (N=227)
Diarrhoea (Gastrointestinal disorders) | 23 (23) | 18 (18)
Nausea (Gastrointestinal disorders) | 11 (11) | 12 (12)
Headache (Nervous system disorders) | 17 (17) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT03198507/SAP_001.pdf
  • Study Protocol (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT03198507/Prot_002.pdf